CLINICAL TRIAL: NCT06721247
Title: Efficacy Of Oral Magnesium Supplementation in Controlled Bronchial Asthma Patients
Brief Title: Oral Intake of Mg in Controlled Asthmatic Patients
Acronym: Mg in asthma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hanaa Sami Hamed, lecturer of chest diseases, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#11325-3/12-2023
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma
MeSH Terms: conditions — Asthma | interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): oral magnesium intake is given to bronchial asthma patients together with the usual asthma medication according to GINA guidelines 2024
  Interventions: Drug: Magnesium; Drug: ICS+LABA
- control group (Placebo Comparator): asthmatic patients who take the usual asthma treatment according to GINA guideline 2024
  Interventions: Drug: ICS+LABA

INTERVENTIONS:
Drug: Magnesium — oral intake of magnesium for asthmatic patients with dose 200 mg per day for one year in addition to usual asthmatic treatment according to GINA guidelines 2024
  Arms: intervention group
Drug: ICS+LABA — inhaled corticosteroids with long acting Beta 2 agonist are given to control group patients twice daily

SUMMARY:
The goal of this clinical trial is to assess the efficacy of oral magnesium supplements in controlled asthmatic patients for proper effective asthma management to reduce frequency of asthma exacerbation & to test the effect of oral magnesium supplementation on improvement of both clinical symptoms and lung functions in patients with bronchial asthma.. The main questions it aims to answer are:

• Can oral supplementation of magnesium play a role in decrease the number of bronchial asthma exacerbations , number of ER visits , number of doctor visits and improve lung function ? Researchers will compare patients on usual treatment according to GINA guidelines 2024 group B and those taking oral magnesium together with the usual group A .

Participants will:

* Take oral magnesium treatment with usual asthma medications according to GINA guidelines (2024) every day for 1year
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their day and night symptoms and the number of times they had activity limitation due to asthma and the number of use reliever.

DETAILED DESCRIPTION:
Asthma is one of the main non-communicable chronic diseases and affects a huge portion of the population. It is a multifactorial disease, classified into several phenotypes, being the allergic the most frequent. The pathophysiological mechanism of asthma involves a Th2-type immune response, with high concentrations of allergen-specific immunoglobulin E, eosinophilia, hyperreactivity and airway remodeling. These mechanisms are orchestrated by intracellular signaling from effector cells, such as lymphocytes and eosinophils. Ion channels play a fundamental role in maintaining the inflammatory response on asthma.The mainstay of management is a beta-agonist and corticosteroids inhaler. However, new investigations into the pathogenesis of the disease are emerging. For example, many reports have observed that low blood levels and low dietary intake of magnesium are factors that possibly contribute to the development of asthma. In addition, low levels of magnesium have been detected in asthmatics compared with non-asthmatics, especially those that have presented to the emergency department with exacerbations.The role of intravenous and inhaled magnesium in the management of acute asthma has been extensively studied and the guidelines are well established. IV or inhaled routes can be used as a last resort for severe, persistent asthma that fails to respond to conventional treatment. Nevertheless, oral magnesium is not included in these guidelines. so on, this study has these objectives : To detect any disturbance in magnesium blood level in patients with controlled bronchial asthma . 2. To compare frequency of asthma exacerbations in asthma controlled patients in patients who will be treated with oral magnesium supplementations and those who will not receive it . 3. To determine if oral magnesium supplementation is an adjunctive from the start for adequate effective control of bronchial asthma. 4. To determine the relationship between oral magnesium supplementation and FEV1 improvement .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Stable controlled asthmatic patients .

Exclusion Criteria:

* Medical conditions and disorders (such as chronic kidney disease, diabetes mellitus, cardiac disease, alcoholism, diarrhea, and pregnancy).
* Any treatment which might affect the absorption or excretion of Mg2+ including digoxin, diuretics, and calcium-containing medications.
* Patients in asthma exacerbations .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
improvement in the degree of asthma control | 6 months to one year
  By using GINA assessment of symptom control and future risk including 1) decrease daytime symptoms of asthma. 2) decrease use of relievers . 3)improvement in daily activities. 4) decrease night awakening due to asthma symptoms .
  By using pulmonary function tests (Spirometer) specially Forced expiratory volume in the first second (FEV1) , any improvement in pulmonary function will be measured .

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No